CLINICAL TRIAL: NCT00094978
Title: Phase I Study of Sequential Depsipeptide/Flavopiridol Infusion for Malignancies Involving Lungs, Esophagus, Pleura, Thymus or Mediastinum
Brief Title: Depsipeptide/Flavopiridol Infusion for Cancers of the Lungs, Esophagus, Pleura, Thymus or Mediastinum
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050010; 05-C-0010; NCT00098644 (obsolete NCT alias)
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2013-05-20

CONDITIONS: Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Mesothelioma
Keywords: Apoptosis; Toxicity; Pharmacokinetic; Gene Induction; Maximally Tolerated Dose; Small Cell Lung Cancer; SCLC; Non-Small Cell Lung Cancer; NSCLC; Esophageal Cancer; Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Mesothelioma; Small Cell Lung Carcinoma; Mesothelioma, Malignant | interventions — Depsipeptides; alvocidib

INTERVENTIONS:
Drug: Depsipeptide
Drug: Flavopiridol (alvocidib)

SUMMARY:
This study will test the safety and effectiveness of two experimental medicines - depsipeptide and flavopiridol - given together to treat cancers of the lung, esophagus, and pleura. It will determine the highest dose that these drugs can safely be given together and will test whether giving them together works better at shrinking tumors than giving either one alone.

Patients 18 years of age and older with cancer of the lung, esophagus, or pleura, or other cancers that have spread to the lungs or pleura may be eligible for this study. Candidates are screened with a medical history and physical examination, blood tests, electrocardiogram (EKG), x-rays and scans, pulmonary function tests, and a tumor biopsy (removal of a small piece of tumor tissue for microscopic examination).

Participants are admitted to the hospital for treatment for approximately 10 days during each 28-day treatment cycle. Depsipeptide is infused through an arm vein or central venous catheter (tube placed in a large vein in the neck or chest) for 4 hours. When this infusion is complete, flavopiridol is infused over 72 hours. The dose of depsipeptide is increased four times over the period of the study with successive groups of patients, and flavopiridol is increased once to determine the maximum safe dose of giving these drugs together.

Blood tests are done before and after each depsipeptide infusion and 3 more times for the next 24 hours, and at various times over 4 days during the flavopiridol infusion to evaluate the effects of the medicines. Samples are also drawn periodically throughout the treatment cycle to evaluate safety. Heart function is monitored with several EKGs before and during the depsipeptide doses. The drug has shown effects on EKG tracings, but does not appear to injure the heart muscle.

Tumor biopsies are done before treatment begins and on the fifth day of the first treatment cycle. The biopsies may be done either in the operating room by passing a tube (bronchoscope) down the throat and into the lungs or in the Radiology Department using a thin needle put through the chest wall into the tumor. For the bronchoscopy, numbing medicine is sprayed into the back of the throat to reduce discomfort, and for the needle biopsy, the skin over the biopsy area is numbed. Optional repeat biopsies may be requested before the start of the second treatment cycle and on day 5 of that cycle. (The repeat biopsies are not required for participation in the study.) At the time of each tumor biopsy, a buccal mucosal biopsy is also done. This involves scraping a tongue depressor along the inside of the mouth to collect cells for examination.

At the end of the first treatment cycle, patients return to NIH for evaluation with a physical examination, blood work, x-rays, and scans of the chest, abdomen, pelvis, and brain. Patients who are not experiencing significant drug side effects are offered a second cycle, exactly like the first. The two cycles complete one course of treatment, after which patients once again return to NIH for evaluation. Additional treatment cycles may be offered to patients whose tumors have shrunk or remained stable with therapy. Patients whose tumors have not responded to therapy or who have developed severe drug side effects are taken off the study.

DETAILED DESCRIPTION:
Background:

In preclinical studies we have demonstrated that the histone deacetylase (HDAC) inhibitor Depsipeptide FR901228 (DP) mediates cell cycle arrest and apoptosis in cultured lung and esophageal cancer, and malignant pleural mesothelioma cells.

We have observed that the cdk inhibitor Flavopiridol (FLA) markedly potentiates Depsipeptide-mediated apoptosis in cultured cancer cells, but not cultured normal epithelial cells.

Patients with advanced malignancies involving lungs, esophagus, or pleura will receive 4-hour Depsipeptide infusion followed by 72-hour FLA infusion using a phase I study design.

Tumor and buccal mucosa biopsies as well as PBMC may be obtained prior to, and after therapy to evaluate gene expression using cDNA array long-oligo and protein lysate array techniques, and determine if sequential DP/FLA mediates apoptosis in target tissues.

Results of these studies may provide the rationale for phase II evaluation of sequential DP/FLA infusion in thoracic oncology patients.

Objectives:<TAB>

Primary objectives:

To define the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of sequential 4 hour Depsipeptide(DP)/72 hour Flavopiridol (FLA)

To evaluate the pharmacokinetics of sequential DP/FLA infusion

Secondary objectives

To analyze gene expression profiles in laser-captured tumor cells, buccal mucosa, and PBMC before and after sequential DP/FLA exposure.

To analyze mcl-1 protein expression and apoptosis in tumor biopsies before and after sequential DP/FLA treatment.

Tertiary objectives:

The development of tissue and serum proteomic techniques to assess treatment response in patients receiving sequential DP/FLA infusions.

Eligibility:

Patients with histologically or cytologically proven primary small cell or non-small cell lung cancers, esophageal cancers, malignant pleural mesotheliomas or chest wall sarcoma, or thymomas are eligible for evaluation. In addition, patients with cancers of nonthoracic origin with metastases to the lungs or pleura, or germ cell tumors refractory to standard therapy are eligible for evaluation.

Patients must have an ECOG performance status of 0 - 2.

Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO greater than the 30 percent predicted, and pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG.

Patients must be 18 years of age or older.

Adequate organ function as evidenced by standard laboratory parameters.

The patient must be willing to sign an informed consent.

Design:<TAB><TAB>

A phase 1 study where patient cohorts will receive escalating doses of Depsipeptide, administered on day 1 and day 21, and a dose of flavopiridol (either 40 mg/m2/d or 50 mg/m2/d) administered on days 1-3, and 21-24 of a 42-day course.

Pharmacokinetics, systemic toxicity, and response to therapy will be recorded.

Two cycles of therapy (one course) will be administered, following which treatment evaluation will be performed using standard clinical criteria.

48 patients will be enrolled over a period of 2-4 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with histologically or cytologically proven small cell or non-small cell lung cancers, esophageal cancers, malignant pleural mesotheliomas chest wall sarcoma, or epithelial thymomas are eligible for evaluation. In addition, patients with cancers of nonthoracic origin with metastases to the lungs, pleura or germ cell tumors refractory to standard therapy are eligible for evaluation.
  2. Chemo naive patients with inoperable lung and esophageal cancers, pleural mesotheliomas, sarcoma, thymomas, as well as tumors of non-thoracic origin with metastasis within the thorax may be eligible for study provided they have been apprised of, and refused potentially effective first line chemotherapy.
  3. Patients with intracranial metastases which have been treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids.
  4. Patients with prior Depsipeptide or Flavopiridol exposure are eligible for study provided they have not experienced dose limiting toxicity at the dose of DP or FLA that they are scheduled to receive.
  5. Patients must have had no chemotherapy, biologic therapy, or radiation therapy for their malignancy for at least 30 days prior to treatment. At least six weeks must elapse between mitomycin C or nitrosourea treatment and DP/FLA therapy. Patients may have received localized radiation therapy to non-target lesions provided that the radiotherapy is completed 14 days prior to commencing therapy, and the patient has recovered from any toxicity.
  6. Patients must have an ECOG performance status of 0 - 2.
  7. Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO greater than the 30% predicted, and pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG.
  8. Patients must be 18 years of age or older due to the unknown effects of HDAC inhibitors and cdk inhibitors during childhood and adolescent development.
  9. Patients must have a platelet count greater than 100,000, an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of less than 1.5 x upper limits of normal, and AST/ALT less than or equal to 1.5 times upper limit of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).
  10. Patients must be aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks. The patient must be willing to sign an informed consent.

EXCLUSION CRITERIA:

1. Patients with limited stage SCLC and operable NSCLC or operable esophageal cancer will be excluded.
2. Patients with potentially treatable pulmonary metastases from lymphomas or germ cell tumors will be excluded.
3. Patients who have received three or more systemic cytotoxic treatment regimens will be excluded due to possible cumulative marrow suppression.
4. Cardiac exclusion criteria, patients with known cardiac abnormalities such as:

   Uncontrolled arrhythmias
   * History of serious ventricular arrhythmias not controlled by coronary artery bypass surgery.
   * Patients with a history of sustained VT, VF, Toursades de Pointes, or cardiac arrest who do not have an automatic implantable cardioverter defibrillator in place.
   * Congenital Long QT syndrome or QTc greater than 480 msec.
   * Patients with Mobitz II second degree block who do not have a pacemaker.
   * Patients with any cardiac arrhythmia requiring anti-arrhythmic medication other than a beta blocker or calcium channel blocker.
   * Patients in whom digitalis cannot be discontinued.

   Decompensated heart failure (NYHA Class II or IV).

   LVEF less than 50% by MUGA scan or echocardiogram.

   Hypertrophic or restrictive cardiomyopathy from prior treatment of other causes and patients with left ventricular hypertrophy.

   Uncontrolled hypertension (i.e. greater than or equal to160/95).

   Myocardial infarction within one year of study.

   Clinically significant active myocardial ischemia on the basis of nuclear imaging or angiography.

   History of coronary artery disease (e.g. angina Canadian Class II-IV or positive stress imaging study).

   Patients with other cardiac disease may be excluded at the discretion of the PI following consultation with cardiology.
5. Co-medication causing QTc prolongation (information at Appendix A and http://georgetowncert.org/gqdrugs_torsades.asp) unless a 5 half-life washout period has elapsed between discontinuing the drug and entering this study.
6. Patients with active intracranial and leptomeningeal metastases, as well as those requiring anticonvulsant medications or steroids to control cerebral edema will be excluded.
7. Patients with life expectancy less than three months will be excluded.
8. Patients with pulmonary embolism or deep venous thrombosis requiring anticoagulation within six months of protocol entry will be excluded.
9. Pregnant patients and nursing mothers will be excluded due to the unknown, potentially harmful effects of HDAC inhibitors and cdk inhibitors on fetal and early childhood development.
10. Patients with active infections will be excluded.
11. Patients with HIV infection will be excluded due to the potential risk of opportunistic infection during DP/FLA-induced myelosuppression and potentially deleterious activation of viral gene expression.
12. Patients will have a screening 12 lead EKG and those patients with left ventricular hypertrophy will not be eligible.
13. Patients who are taking hydrochlorothiazide (HCTZ) will have this agent stopped or switched to a potassium-conserving combination (e.g. Maxide or Dyazide) or other antihypertensive agent. Patients, who cannot have the agent stopped or switched to a potassium-conserving combination or other antihypertensive agent, will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-10-25; Primary Completion 2013-05-20 (Actual); Study Completion 2013-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Otterson GA, Khleif SN, Chen W, Coxon AB, Kaye FJ. CDKN2 gene silencing in lung cancer by DNA hypermethylation and kinetics of p16INK4 protein induction by 5-aza 2'deoxycytidine. Oncogene. 1995 Sep 21;11(6):1211-6. PMID 7566983
- [Background] Baylin SB, Esteller M, Rountree MR, Bachman KE, Schuebel K, Herman JG. Aberrant patterns of DNA methylation, chromatin formation and gene expression in cancer. Hum Mol Genet. 2001 Apr;10(7):687-92. doi: 10.1093/hmg/10.7.687. PMID 11257100
- [Background] Wang C, Fu M, Mani S, Wadler S, Senderowicz AM, Pestell RG. Histone acetylation and the cell-cycle in cancer. Front Biosci. 2001 Apr 1;6:D610-29. doi: 10.2741/1wang1. PMID 11282573